CLINICAL TRIAL: NCT03160027
Title: Examining the Impact of Photobiomodulation (PBM) on Brain Function in Dementia
Brief Title: Photobiomodulation for Improving Brain Function in Dementia (PBM Dementia)
Acronym: PBM Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-21406
Record Dates: First submitted 2017-05-16; First posted 2017-05-19 (Actual); Results first posted 2019-08-20 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Dementia, Alzheimer Type
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Participants randomized to the "Immediate PBM treatment" group will receive 12 weeks of PBM, delivered with the Vielight Neuro device, for 12 weeks, once every other day (e.g., Mon, Wed, Fri), undergo behavioral assessments at baseline, weeks 6 and 12, and undergo 3 Tesla MRI at baseline and week 12.
  Participants randomized to the "Delayed PBM treatment" group will maintain their usual activities for 12 weeks, undergo behavioral assessments at baseline, weeks 6 and 12, and undergo 3 Tesla MRI at baseline and week 12. After the week 12 behavioral and MRI assessments, participants in this group will receive 12 weeks of PBM, delivered with the Vielight Neuro device, for 12 weeks, once every other day (e.g., Mon, Wed, Fri), undergo behavioral assessments at weeks 18 and 24.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Immediate PBM treatment (Experimental): This arm will receive photobiomodulation (PBM), delivered with the Vielight Gamma device, once every other day (e.g., Mon, Wed, Fri) for 20 minutes (the device automatically shuts itself off after 20 minutes) for 12 weeks.
  Interventions: Device: Vielight Neuro Gamma
- Delayed PBM treatment (No Intervention): This arm will maintain usual activities for 12 weeks. After the week 12 psychometric and MRI assessment, this arm will receive PBM, delivered with the Vielight Gamma device, once every other day (e.g., Mon, Wed, Fri) for 20 minutes (the device automatically shuts itself off after 20 minutes) for 12 weeks.

INTERVENTIONS:
Device: Vielight Neuro Gamma — The Vielight Neuro Gamma is headset that delivers transcranial (through the scalp and skull) and intranasal (through the nose) near infrared (NIR) light. The device is engineered for increased efficacy and easy domestic use for comprehensive brain photobiomodulation (PBM). The NIR lights are pulsed at a 40 Hz rate, which correlates with electroencephalogram (EEG) gamma brain wave entrainment.
  Arms: Immediate PBM treatment

SUMMARY:
A recent study (Saltmarche et al., 21017) examined the effects of photobiomodulation (PBM), a kind of light therapy that uses red or near-infrared light to heal and protect tissue that has either been injured, is degenerating, or else is at risk of dying, in 5 older adults with dementia. After 12 weeks of PBM treatments, delivered with a commercially available, wearable device, the patients with mild to moderately severe dementia showed improvements on the Mini-mental State Exam (MMSE, p<0.003) and Alzheimer's Disease Assessment Scale-cognitive, ADAS-cog, p<0.03). The caregivers, who kept daily journals of their experiences during the 12 weeks of PBM treatment, reported better sleep, fewer angry outbursts, decreased anxiety and wandering in their loved-ones with dementia. The goals of this trial are to: (1) replicate this finding in a larger group of individuals with dementia and (2) to examine the underling brain mechanisms behind the changes in cognitive function.

DETAILED DESCRIPTION:
Photobiomodulation (PBM) describes a kind of light therapy that uses red or near-infrared light to stimulate, heal, regenerate, and protect tissue that has either been injured, is degenerating, or else is at risk of dying. Human cadaver studies have shown near-infrared wavelengths can penetrate 40-50 mm through the scalp and skull. Saltmarche et al. (2017) recently reported that 12-weeks of transcranial treatment with a commercially available PBM device (i.e., the Vielight "Neuro ") benefits cognitive function in patients with mild-to-moderately severe dementia. Specifically, Saltmarche et al. reported improvements on the Mini Mental State Examination (MMSE, p< 0.003) and Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog, p< 0.03) in 5 dementia patients after 12-weeks of PBM treatment.

The first aim of this trial is to replicate Saltmarche et al' s findings that the effects of 12-weeks of PBM treatment can improve cognitive function in older adults with dementia. Because the Vielight Neuro device targets nodes of the default mode network (DMN), which is dysregulated in Alzheimer's disease (AD), the second aim of this pilot study is to investigate whether 12 weeks of PBM therapy with the Vielight Neuro device improves DMN connectivity in older adults with dementia. Finally, because there is suggestive evidence that PBM therapy enhances blood flow, the third aim of the trial is to examine whether 12-weeks of PBM therapy improves cerebral blood flow (CBF) in older adults with dementia. The trial will also explore the effects of PBM treatment on quality of life in older adults with dementia and on caregiver burden.

Ten older adults with dementia (i.e., the primary study participants, PP) and their caregivers (CG) will be enrolled in a randomized, wait-list control trial. Five PPs will be randomized to the "immediate" PBM treatment group after the baseline psychometric and MRI assessments. Five PP will be randomized to a "delayed" PBM treatment group that will not receive PBM treatment with the Vielight Neuro device until after the 12 week psychometric and MRI assessments.

Neuroimaging measures will be assessed in all PPs at baseline and week 12. Cognitive function and quality of life will be assessed in all PPs at baseline, weeks 6 and 12. Caregivers (CGs) will be asked to fill out questionnaires Caregivers (CGs) will be asked to fill out questionnaires about caregiver burden, positive aspects of care giving, depressive symptomology, and dementia-related behaviors in the PP at baseline, weeks 6 and 12.

PPs randomized to the "immediate" PBM treatment group will receive PBM with the Vielight Neuro device once a day, every other day (e.g., Mon, Wed, Fri) for 12 weeks. PPs randomized to the "delayed" PBM treatment group will keep doing their usual activities for 12 weeks. After the 12 week psychometric and MRI assessments, PPs randomized to the "delayed" PBM treatment group will receive PBM with the Vielight Neuro device once a day, every other day (e.g., Mon, Wed, Fri) for 12 weeks. PPs randomized to the "delayed" PBM treatment group will undergo additional psychometric assessment at weeks 18 and 24. CGs of PPs randomized to the "delayed" PBM treatment group will be asked to fill out additional questionnaires about caregiver burden, positive aspects of care giving, depressive symptomology, and dementia-related behaviors in the PP at baseline, weeks 18 and 24.

ELIGIBILITY:
Inclusion Criteria:

For primary study participants (i.e., individuals with dementia):

age > 50 years a diagnosis of dementia (preferably AD) by their neurologist English language fluency, legally authorized representative consent no contraindications for MRI MMSE > 11

Inclusion criteria for caregivers:

current provision of care to primary participant with dementia ability to answer questions about the primary participant's behaviors, quality of life, and their own level of stress.

Exclusion Criteria:

For primary study participants (i.e., individuals with dementia):

lack of assent to study procedures contraindications for MRI (i.e., pacemakers, metal implants, claustrophobia) terminal illness (i.e., life expectancy < 1 year) started dementia medication (i.e., cholinesterase inhibitor or memantine) in the past 3 months or planning to start new dementia medication current participation in another research study that could potentially confound current study (e.g., medication or behavioral intervention) MMSE < 11.

Exclusion criteria for caregivers:

major neurological or psychiatric condition terminal illness evidence of cognitive impairment inability to consent to study procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda L Chao, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco Veterans Affairs Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate PBM Treatment - Patients: This arm will receive photobiomodulation (PBM), delivered with the Vielight Gamma device, once every other day (e.g., Mon, Wed, Fri) for 20 minutes (the device automatically shuts itself off after 20 minutes) for 12 weeks.
  Vielight Neuro Gamma: The Vielight Neuro Gamma is headset that delivers transcranial (through the scalp and skull) and intranasal (through the nose) near infrared (NIR) light. The device is engineered for increased efficacy and easy domestic use for comprehensive brain photobiomodulation (PBM). The NIR lights are pulsed at a 40 Hz rate, which correlates with electroencephalogram (EEG) gamma brain wave entrainment.
- Delayed PBM Treatment - Patients: This arm will maintain usual activities for 12 weeks. After the week 12 psychometric and MRI assessment, this arm will receive PBM, delivered with the Vielight Gamma device, once every other day (e.g., Mon, Wed, Fri) for 20 minutes (the device automatically shuts itself off after 20 minutes) for 12 weeks.
- Immediate PBM Treatment - Caregivers: This arm consists of the caregivers of patients who will receive photobiomodulation (PBM), delivered with the Vielight Gamma device, once every other day (e.g., Mon, Wed, Fri) for 20 minutes.
- Delayed PBM Treatment - Caregivers: This arm consists of caregivers of patients who will maintain usual activities for 12 weeks.
Period: Overall Study
Arm/Group | Immediate PBM Treatment - Patients | Delayed PBM Treatment - Patients | Immediate PBM Treatment - Caregivers | Delayed PBM Treatment - Caregivers
Started | 6 | 4 | 6 | 4
Completed | 6 | 4 | 6 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients + Study Partner randomized to Immediate or Delayed PBM treatment
Groups:
- Immediate PBM Treatment - Patient: This arm will receive photobiomodulation (PBM), delivered with the Vielight Gamma device, once every other day (e.g., Mon, Wed, Fri) for 20 minutes (the device automatically shuts itself off after 20 minutes) for 12 weeks.
  Vielight Neuro Gamma: The Vielight Neuro Gamma is headset that delivers transcranial (through the scalp and skull) and intranasal (through the nose) near infrared (NIR) light. The device is engineered for increased efficacy and easy domestic use for comprehensive brain photobiomodulation (PBM). The NIR lights are pulsed at a 40 Hz rate, which correlates with electroencephalogram (EEG) gamma brain wave entrainment.
- Immediate PBM Treatment - Study Partner: This arm will help administer photobiomodulation (PBM), delivered with the Vielight Gamma device, once every other day (e.g., Mon, Wed, Fri) for 20 minutes (the device automatically shuts itself off after 20 minutes) for 12 weeks to the patient.
- Delayed PBM Treatment - Patient: This arm will maintain usual activities for 12 weeks. After the week 12 psychometric and MRI assessment, this arm will receive PBM, delivered with the Vielight Gamma device, once every other day (e.g., Mon, Wed, Fri) for 20 minutes (the device automatically shuts itself off after 20 minutes) for 12 weeks.
- Delayed PBM Treatment - Study Partner: This arm will maintain usual activities for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Immediate PBM Treatment - Patient | Immediate PBM Treatment - Study Partner | Delayed PBM Treatment - Patient | Delayed PBM Treatment - Study Partner | Total
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 78.3 (10.2) | 75.0 (10.8) | 79.0 (5.9) | 50.5 (14.3) | 78.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 3 | 11
  Male | 3 | 3 | 2 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 4 | 4 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 4 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Alzheimer's Disease Assessment Scale-cognitive Subscale (ADAS-cog)
Description: The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog) test is one of the most frequently used tests to measure cognition in research studies and clinical trials for new drugs and other interventions. It consists of 11 tasks measuring the disturbances of memory, language, praxis (e.g., ability to conceptualize, plan, and execute the complex sequences of motor actions), attention and other cognitive abilities which are often referred to as the core symptoms of AD. The ADAS-cog score is based on the number of errors made in each item. Total score ranges from 0 to 70. A score of 70 represents the most severe impairment. A score of 0 represents the least impairment.
  This outcome is a change score, derived by subtracting Baseline ADAS-cog score from Week 12 ADAS-cog score.
Time Frame: change from baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on the ADAS-cog scale
Groups:
- Delayed PBM After 12 Weeks of PBM: Delayed PBM participants who opted to undergo 12 weeks of PBM treatments after 12 weeks of Usual Care
Arm/Group | Immediate PBM Treatment | Delayed PBM Treatment | Delayed PBM After 12 Weeks of PBM
Number analyzed (Participants) | 4 | 4 | 3
units on the ADAS-cog scale | 5.8 (1.7) | -7.2 (5.8) | 4.8 (2.2)

2. Primary Outcome: Change in Clock-drawing Test
Description: The clock-drawing test is used for screening for cognitive impairment and dementia and as a measure of spatial dysfunction and neglect. The score ranges from 0 (none correct) to 5 (all correct). A score greater than or equal to 4 is considered "normal" The outcome is a change score: Baseline - Week 12 score. Or Week 12 - Week 24 for Delayed PBM participants who opted to undergo 12 weeks of PBM treatments after 12 weeks of Usual Care. A negative change score = improvement; a positive change score = decline.
Time Frame: change from baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on clock-drawing test score
Groups:
- Delayed PBM After 12 Weeks of PBM: Delayed PBM patients who opted to undergo 12 weeks of
Arm/Group | Immediate PBM Treatment | Delayed PBM Treatment | Delayed PBM After 12 Weeks of PBM
Number analyzed (Participants) | 4 | 4 | 3
units on clock-drawing test score | 0.3 (1.3) | 0.5 (1.0) | 0 (0)

3. Primary Outcome: Change in Default Mode Network (DMN) Functional Connectivity
Description: The DMN is a network of interacting brain regions known to have activity highly correlated with each other and distinct from other networks in the brain. This outcome consists of the strength of the connection between the posterior cingulate cortex (PCC), a hub of the DMN, and the left (L) and right (R) lateral parietal cortex (LP) at baseline and at Week 12. Studies in patients with Alzheimer's disease (AD) suggest there is diminished connectivity between nodes of the DMN in AD. Therefore increased connectivity between nodes of the DMN from baseline to Week 12 (or higher T-scores of the connection) indicate better outcomes. The measure type of "number" for this assessment is the T-score that was calculated for each "group".
Time Frame: change from baseline to 12 weeks
Measure: Number; unit: T-score
Arm/Group | Immediate PBM Treatment | Delayed PBM Treatment
Number analyzed (Participants) | 4 | 4
T-score
  strength of connection bet. PCC & LLP at baseline | 4.25 | 6.88
  strength of connection bet. PCC & LLP at Week 12 | 14.15 | 3.86
  strength of connection bet. PCC & RLP at baseline | 3.98 | 8.34
  strength of connection bet. PCC & RLP at Week 12 | 11.17 | 5.04

4. Primary Outcome: Change in Arterial Spin Labeled (ASL) Perfusion MRI Measure
Description: This outcome consists of measures of blood flow to the brain at baseline and at Week 12. Total perfusion values were derived by averaging across the superior frontal, superior parietal, and supramarginal regions of interest (ROI), based on the location of the transcranial LED clusters. The perfusion values were normalized to the precentral gyrus (i.e., motor cortex) perfusion .
Time Frame: change from baseline to 12 weeks
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Immediate PBM Treatment | Delayed PBM Treatment
Number analyzed (Participants) | 4 | 4
ratio
  Baseline total perfusion | 0.89 (0.11) | 1.20 (0.11)
  Week 12 total perfusion | 1.22 (0.16) | 0.91 (0.16)

5. Primary Outcome: Change in Quality of Life Scale in Alzheimer's Disease (QOL-AD)
Description: The QOL-AD is a standard quality of life measure that asks parallel questions of affected individuals and their caregivers. Current quality of life is rated as poor (1 point), fair (2 points), good (3 points) or excellent (4 points) in 13 areas: physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores around the house, ability to do things for fun, money, and life as a whole. Score range from 0 (worse quality of life) to 52 (best quality of life)
  This outcome is a change score, derived by subtracting Baseline from Week 12 scores (or Week 12 - Week 24) for Delayed PBM participants who chose to undergo 12 weeks of PBM after 12 weeks of Usual Care). A higher change score = decline in perceived quality of life. A lower or negative change score = improved perceived quality of life.
Time Frame: change from baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on QOL-AD score
Groups:
- Delayed PBM After 12 Weeks of PBM: Delayed PBM participants who chose to undergo 12 weeks of PBM treatments after 12 weeks of Usual Care
Arm/Group | Immediate PBM Treatment | Delayed PBM Treatment | Delayed PBM After 12 Weeks of PBM
Number analyzed (Participants) | 4 | 4 | 3
units on QOL-AD score | 1.5 (3.7) | -0.3 (3.6) | 3 (3.5)

6. Secondary Outcome: Change in QOL-AD From the Caregiver's Perspective About the Individual With Dementia
Description: This outcome is a change in the quality of life of the individual with dementia from the caregiver's perspective. Scores range from 52 (best possible perceived quality of life) to 0 (worse possible perceived quality of life). A positive or larger change score = decreased quality of life. A negative or smaller change score = improved quality of life.
Time Frame: change from baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on QOL-AD score
Arm/Group | Immediate PBM Treatment | Delayed PBM Treatment | Delayed PBM After 12 Weeks of PBM
Number analyzed (Participants) | 4 | 4 | 3
units on QOL-AD score | 1.8 (5.0) | 3.8 (3.8) | -2.3 (1.5)

7. Secondary Outcome: Change in Caregiver Burden Inventory (CBI).
Description: The CBI is a standard measure that includes 24 items and 5 domains. Caregivers are asked to rate how often each statement describes their feelings (never, rarely, sometimes, quite frequently, nearly always). The total score may range from 0 to 96 with higher scores reflecting greater feelings of burden. This outcome is a change score: Baseline CBI score - Week 12 CBI score. A positive (or larger) change score = decrease in caregiver burden. A negative (or smaller) chance score = increase in caregiver burden.
Time Frame: change from baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on the CBI scale
Arm/Group | Immediate PBM Treatment | Delayed PBM Treatment | Delayed PBM After 12 Weeks of PBM
Number analyzed (Participants) | 4 | 4 | 3
units on the CBI scale | 12.0 (20.7) | -7.8 (9.6) | -2.5 (3.4)

8. Secondary Outcome: Change in Neuropsychiatric Inventory (NPI)
Description: The NPI assesses the frequency and severity of 12 common dementia-related behaviors (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep and appetite/eating). It is a questionnaire completed by the caregiver about the individual with dementia. The total NPI score ranges from 0 to 144. A higher the total NPI score signifies more numerous, frequent, and/or more severe dementia-related behaviors.
  This outcome is a change score: Baseline NPI score - Week 12 NPI score. (or Week 12 - Week 24 for Delayed PBM participants who opted to undergo PBM treatments) A positive (or larger) change score = decrease in the number and/or severity of dementia-related behaviors. A negative (or smaller) change score = increase in the number and/or severity of dementia-related behaviors.
Time Frame: change from baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on CBI scale
Groups:
- Delayed PBM After 12 Weeks of PBM: Delayed PBM participants who opted to undergo 12 weeks fo PBM treatments after 12 weeks of Usual Care
Arm/Group | Immediate PBM Treatment | Delayed PBM Treatment | Delayed PBM After 12 Weeks of PBM
Number analyzed (Participants) | 4 | 4 | 3
units on CBI scale | 17.8 (24.4) | -2.0 (4.5) | 6.7 (4.5)

9. Secondary Outcome: Change in Positive Aspects of Caregiving Scale
Description: The Positive Aspects of Caregiving Scale is a standard measure that asks caregivers to rate their agreement/disagreement with 11 statements about positive aspects of caregiving on a 5-point likert scale (disagree a lot ... agree a lot). Scores can range from 11 (few positive aspects of providing care for someone with dementia) to 55 (many positive aspects of providing care for someone with dementia).
  This outcome is a change score: Week 12 score - baseline score. A larger (or positive) change score = increase in positive aspects of caregiving. A negative (or smaller) change score = decrease in positive aspects of caregiving.
Time Frame: change from baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on Positive Aspects of Caregiving
Arm/Group | Immediate PBM Treatment | Delayed PBM Treatment | Delayed PBM After 12 Weeks of PBM
Number analyzed (Participants) | 4 | 4 | 3
units on Positive Aspects of Caregiving | 0.3 (3.7) | 0.0 (3.2) | -0.3 (5.1)

10. Secondary Outcome: Change in Geriatric Depression Scale (GDS) - Short Form in the Caregivers
Description: The GDS-short form is a 15-item yes/no scale that measures depressive symptoms in older individuals. Scores range from 0-15. Higher scores reflect the presence of more depressive symptoms. A score of 0-5 is normal; a score > 5 suggests depression; a score ≥ 10 is strong indicator of depression.
  This outcome is a change score: Baseline GDS score - Week 12 GDS score. In participants randomized Delayed PBM treatment who opt to undergo PBM treatments after 12 weeks of Usual Care, Week 12 GDS score - Week 24 GDS score. A positive (or larger) change score = decrease in depressive symptoms in caregivers. A negative (or smaller) change score = increase in depressive symptoms in caregivers.
Time Frame: change from baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on the Geriatric Depression Scale
Arm/Group | Immediate PBM Treatment | Delayed PBM Treatment | Delayed PBM After 12 Weeks of PBM
Number analyzed (Participants) | 4 | 4 | 3
units on the Geriatric Depression Scale | -0.3 (1.0) | 0.0 (0.8) | -0.3 (1)

ADVERSE EVENTS:
Time Frame: 24 weeks (12 weeks for all participants; adverse events were assessed an additional 12 weeks for Delayed PBM participants who chose to undergo 12 weeks of PBM treatments after 12 weeks of Usual Care)
Groups:
- Delayed PBM Participants Who Underwent PBM Treatment After: This arm consists of Delayed PBM participants who opt to undergo 12 weeks of PBM treatments after maintaining usual activities for 12 weeks. After the Week 12 psychometric and MRI assessments, participants arm will receive PBM, delivered with the Vielight Gamma device, once every other day (e.g., Mon, Wed, Fri) for 20 minutes (the device automatically shuts itself off after 20 minutes) for 12 weeks.
Arm/Group | Immediate PBM Treatment | Delayed PBM Treatment | Delayed PBM Participants Who Underwent PBM Treatment After
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
(1) small sample size, (2) absence of a sham-control group, (3) the patients' diagnoses of dementia were not independently confirmed by a neurologist, and (4) adherence to the PBM treatment protocol was solely monitored in home treatment diaries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT03160027/Prot_SAP_000.pdf